CLINICAL TRIAL: NCT04365023
Title: Epidemiological Study of the Therapeutic Management of Well-differentiated Grade 3 (WHO Classification) Neuroendocrine Digestive Tumors From the Prospective Data of the French Neuroendocrine Tumors Registry (GTE)
Brief Title: Cohort of Well-differentiated Grade 3 Neuroendocrine Digestive Tumors
Acronym: TNE-bien-DIF
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: NI18009HLJ; 2019-A00404-53 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2020-04-25; First posted 2020-04-28 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Neuroendocrine Tumors
Keywords: Neuroendocrine Tumors; Epidemiology
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Well-differentiated grade 3 gastrointestinal neuroendocrine tumors patients who receive first line platinum based chemotherapy
  Interventions: Drug: platinum chemotherapy
- 2: Well-differentiated grade 3 gastrointestinal neuroendocrine tumors patients who receive receiving first line non-platinum chemotherapy

INTERVENTIONS:
Drug: platinum chemotherapy — First line platinum chemotherapy
  Groups: 1

SUMMARY:
The purpose of this study is to analyse clinical data of well-differentiated grade 3 digestive neuroendocrine tumors. These rare tumors may have a different disease evolution, response to chemotherapy and prognostic.

DETAILED DESCRIPTION:
Digestive neuroendocrine tumors are rare tumors and cell differentiation is a major prognostic marker of neuroendocrine tumors.

The 2010 WHO Classification defined three groups of tumor according to the combination of the morphological characteristics and the mitotic index and/or the Ki-67 index: Grade 1 and 2 corresponded to well differentiated neuroendocrine tumors whereas grade 3 corresponded to poorly differentiated lesions entitled neuroendocrine carcinomas (NEC). It was assumed that no well-differentiated neuroendocrine tumor with a mitotic- or a Ki-67- index above 20% existed.

Recently, a proportion of neuroendocrine tumors corresponding to grade 3 neuroendocrine tumors with a proliferation- or Ki-67 index > 20% and with a well-differentiated morphology have been identified. This entity has been partially explored and may have a different survival than grade 3 NEC. Furthermore, targeted therapies, and used in pancreatic neuroendocrine tumors have not been assessed in this case.

The TENpath network is a pathological network whose goal is the systematic reading of all diagnosed cases of neuroendocrine tumors. As part of this network, nearly 3.000 neuroendocrine tumors were reviewed by pathologist experts. Of all the reviewed tumors, 167 were identified as well-differentiated grade 3 neuroendocrine tumors, observed Ki-67(5.6%) confirming the existence of this entity.

Treatment and follow-up of well-differentiated grade 3 tumors are not consensus-based and recommendations are exclusively based on experts' opinions. The purpose of this study is to define the characterization of this entity and evaluate the efficacy of chemotherapy on well-differentiated grade 3 digestive neuroendocrine tumors identified from the TENpath network.

ELIGIBILITY:
Inclusion Criteria:

* Well-differentiated grade 3 neuroendocrine digestive tumors
* Patient of 18 years old and more

Exclusion Criteria:

* Patient opposed to data collection as part of the study
* Digestive neuroendocrine tumors Grade 1-2
* Grade 3 poorly differentiated digestive neuroendocrine tumors
* Malignant disease diagnosed in the last 5 years (except basal cell of the skin and in situ cervical carcinoma)
* Other non-digestive neuroendocrine tumors
* Mixed neuroendocrine non neuroendocrine neoplasm

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: digestive tumors recorded in the national registry of endocrine tumors (GTE) and the TENpath registry
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Title : Overall survival | 12 months
  To compare the median of overall survival of Well-differentiated grade 3 gastrointestinal neuroendocrine tumors patients who receive first line platinum based chemotherapy versus patients receiving first line non-platinum chemotherapy

SECONDARY OUTCOMES:
Objective response rate | 12 months
Progression Free Survival | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Romain CORIAT, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Gastroenterology and digestive oncology unit - Cochin hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No